CLINICAL TRIAL: NCT01727973
Title: Efficacy of Subantimicrobial Dose Doxycycline for Moderate to Severe and Active Graves' Orbitopathy: a Prospective, Uncontrolled Pilot Study
Brief Title: Efficacy of Subantimicrobial Dose Doxycycline for Moderate to Severe and Active Graves' Orbitopathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Dan Liang, MD, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO-DOXY-1
Record Dates: First submitted 2012-11-12; First posted 2012-11-16 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Graves Ophthalmopathy; Graves Disease; Eye Diseases; Thyroid Diseases; Endocrine System Diseases; Eye Diseases, Hereditary; Hyperthyroidism; Autoimmune Diseases; Immune System Diseases
Keywords: Graves' orbitopathy; Graves´ ophthalmopathy; Thyroid eye disease; Thyroid-associated ophthalmopathy; Doxycycline; EUGOGO; CAS
MeSH Terms: conditions — Graves Ophthalmopathy; Graves Disease; Eye Diseases; Thyroid Diseases; Endocrine System Diseases; Eye Diseases, Hereditary; Hyperthyroidism; Autoimmune Diseases; Immune System Diseases | interventions — Doxycycline; sulfadiazine, tetroxoprim drug combination; Chlortetracycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Doxycycline (Experimental): Tablets Doxycycline 50 mg PO per day for 12 weeks
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Doxycycline — Tab. Doxycycline 50 mg PO per day for 12 weeks
  Other Names: Dolotard; Tibirox; Biomycin

SUMMARY:
The aim of this study is to evaluate the effects of subantimicrobial dose doxycycline (50 mg/d), administered for 12 wk, for patients with active moderate-severe Graves' Orbitopathy (GO).

DETAILED DESCRIPTION:
Graves'orbitopathy is an autoimmune disease characterised by an inflammatory phase followed by fibrosis. Surgery to correct eyelid swelling, proptosis, and diplopia is effective, but can not be done until the inflammatory phase has passed. To arrest the inflammatory phase, several types of immunosuppressive treatments have been investigated. Corticosteroids are the first-choice immunosuppressive treatment, but they often cause severe side-effects.

Subantimicrobial dose doxycycline posses known anti-inflammatory effects that are separate from their antibacterial mode of action. This mode of action has lead to the routine use of subantimicrobial dose doxycycline for rosacea, periodontitis and multiple sclerosis.

We propose to test the effect of subantimicrobial dose doxycycline for non-sight threatening, moderate-severe, inflammatory GO.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Graves' Orbitopathy
* Moderate-severe GO According to EUGOGO statements, patients with moderate-severe GO usually have any one or more of the following：moderate or severe soft tissue involvement, exophthalmos≥3mm above normal for race and gender, inconstant, or constant diplopia.
* Clinical activity score ≥ 3
* Being euthyroid for at least 1 month before the date of inclusion
* Must be able to swallow tablets
* Written informed consent is obtained

Exclusion Criteria:

* Mild Graves' Orbitopathy
* Sight-threatening Graves' Orbitopathy
* Clinical activity score < 3
* Previous treatment for GO Oral steroids, intravenous steroids, radiotherapy
* Pregnant females as determined by positive (serum or urine) Human chorionic gonadotropin (hCG) test at screening or prior to dosing, or lactating females
* Uncontrolled diabetes or hypertension
* History of mental / psychiatric disorder
* Hepatic dysfunction (Albumin (Alb),Aspartate Transaminase (AST), Alanine Aminotransferase (ALT) and Alkaline phosphates levels must be within normal range for eligibility)
* Renal impairment (Urea and Creatinine levels must be within normal range)
* Doxycycline allergy or intolerance

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2012-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
• Treatment response | 24 weeks
  As definition of treatment response, we used the major and minor criteria . Three major criteria were: improvement in diplopia grade (disappearance or change in grade); improvement of ≥8 degrees in any direction of eye movements; reduction of three points or more in CAS. Four minor criteria were: reduction of 2 mm or more in eyelid aperture; reduction of 2 mm or more in proptosis; improvement in grade of soft tissue swelling; decrease in CAS by at least two points. A successful response was defined as an improvement in one or more major criteria or in two minor criteria, in absence of deterioration of any criterion in that observed eye. Deterioration was defined as occurrence of DON, and/or worsening of soft tissue swelling, and/or worsening of diplopia, and/or an increase of ≥2 mm in lid aperture, and/or an increase of ≥2 mm in proptosis, and/or a decrease of ≥8 degrees in duction. No success was defined if there was no change or the changes did not reach the success criteria.

SECONDARY OUTCOMES:
Safety and tolerability as assessed by adverse events, vital signs | 24 weeks
Graves' orbitopathy-Specific Quality of Life (GO-QoL) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dan Liang, MD, Principal Investigator — Zhongsh Ophthalmic Center
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Lin M, Mao Y, Ai S, Liu G, Zhang J, Yan J, Yang H, Li A, Zou Y, Liang D. Efficacy of Subantimicrobial Dose Doxycycline for Moderate-to-Severe and Active Graves' Orbitopathy. Int J Endocrinol. 2015;2015:285698. doi: 10.1155/2015/285698. Epub 2015 Jun 29. PMID 26221138
- See also: Genetics Home Reference related topics: Lenz microphthalmia syndrome oculofaciocardiodental syndrome Peters plus syndrome — http://ghr.nlm.nih.gov/
- See also: MedlinePlus related topics: Antibiotics Eye Diseases Thyroid Diseases — http://www.nlm.nih.gov/medlineplus
- See also: Drug Information available for: Doxycycline Dolotard Tibirox Biomycin — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp
- See also: U.S. FDA Resources — http://www.clinicaltrials.gov/ct2/info/fdalinks